CLINICAL TRIAL: NCT02810964
Title: A Double-Blind Placebo-Controlled Trial of a Sulforaphane Nutraceutical to Reduce the Symptoms of Schizophrenia
Brief Title: Sulforaphane to Reduce Symptoms of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Responsible Party: Principal Investigator, Faith Dickerson, Principal Investigator, Stanley Research Program, Sheppard Pratt Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMRI/SPHS: 2016-01
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Sulforaphane; Sulforaphane supplement
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulforaphane Nutraceutical (Experimental): The sulforaphane nutraceutical contains inactive glucoraphanin, a glucosinolate from broccoli seeds, and myrosinase from broccoli sprouts. The ingestion of this compound leads to the hydrolysis of glucoraphanin, the generation of sulforaphane within the gastrointestinal (GI) tract, and the subsequent systemic absorption of the sulforaphane. The dose per tablet is 16 mg of glucoraphanin or 37 µmol; 6 tablets per day should yield about 100 µmol of sulforaphane. The tablets, which will be swallowed, are provided as .375 punch size, round concave tablets. In this arm, the participant will take 6 tablets of the sulforaphane nutraceutical daily for 16 weeks after a 2-week placebo run-in.
  Interventions: Drug: Sulforaphane Nutraceutical
- Identical-appearing Placebo (Placebo Comparator): The inert compound placebo looks identical to the sulforaphane nutraceutical. In this arm, the participant will take 6 tablets of the placebo daily for 16 weeks after a 2-week placebo run-in.
  Interventions: Drug: Identical-appearing Placebo

INTERVENTIONS:
Drug: Sulforaphane Nutraceutical — Sulforaphane Nutraceutical 6 tablets by mouth daily
  Other Names: Avmacol®
  Arms: Sulforaphane Nutraceutical
Drug: Identical-appearing Placebo — Identical-appearing Placebo 6 tablets by mouth daily
  Arms: Identical-appearing Placebo

SUMMARY:
The purpose of this study is to determine if taking a sulforaphane nutraceutical versus a placebo will reduce symptoms of schizophrenia when used in addition to standard antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* Capacity for written informed consent
* Age 18-65 years, inclusive
* Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder as determined by the Structured Clinical Interview for DSM-5 Disorders (SCID-5)
* Currently an outpatient at time of screening
* Residual psychotic symptoms of at least moderate severity as evidenced by a Positive and Negative Syndrome Scale (PANSS) total score of 60 or higher AND one or more of the following: one or more PANSS positive symptom scores of 4 or higher; OR containing at least three positive or negative items with scores of 3 or higher at the screening visit
* Receiving antipsychotic medication for at least 8 weeks prior to enrolling in the study with no antipsychotic medication changes within the previous 21 days from visit 2 (week 0)
* Conformance to PORT Treatment Recommendation about Maintenance Antipsychotic Medication Dose
* Proficient in the English language
* Participated previously in one of our screening studies

Exclusion Criteria:

* Any clinically significant or unstable medical disorder as determined by the principal investigator and/or the study physician (e.g., HIV infection or other immunodeficiency condition (such as receiving chemotherapy), uncontrolled diabetes, congestive heart failure)
* DSM-5 diagnosis of intellectual disability or comparable diagnoses determined by previous versions of the DSM
* DSM-5 diagnosis of a moderate or severe substance use disorder, except for caffeine or tobacco, within the last three months prior to the screening visit. If the patient has a positive drug toxicity screen at the time of visit 1 (screening), further evaluation by the investigator will be done of the substance use to determine eligibility.
* Any current use of a broccoli supplement (e.g., Avmacol® or other health food broccoli supplement)
* Participated in any investigational drug trial in the past 30 days prior to the screening visit
* Pregnant, planning to become pregnant, or breastfeeding during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Dickerson, PhD, MPH, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppart Pratt Health System, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, symptom, and cognitive data will be shared with the National Database for Clinical Trials Related to Mental Illness (NDCT). Access may be obtained through an approved application with the NDCT.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled n=64 participants drawn from rehabilitation and treatment programs in Central Maryland. Dates of recruitment: February 2017 - June 2019.
Pre-assignment Details: We used a 2 week single-blind placebo phase for all participants prior to randomization. This placebo run-in was followed by the 16 week double-blind treatment phase.
Groups:
- Sulforaphane Nutraceutical: Sulforaphane nutraceutical 6 tablets by mouth daily for 16 weeks
- Identical-appearing Placebo: Identical-appearing placebo 6 tablets by mouth daily for 16 weeks
Period: Placebo Run-In Phase (2 Weeks)
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0
Period: Double-Blind Treatment Phase (16 Weeks)
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Started | 32 | 32
Completed | 29 | 29
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Relocation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.3) | 45.8 (11.7) | 44.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 24 | 25 | 49
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 18 | 16 | 34
  African American | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Score From the Start to the End of the Double-blind Treatment Phase
Description: The Positive and Negative Syndrome Scale (PANSS) measures psychiatric symptomatology, especially related to psychosis. The complete PANSS contains ratings for 30 symptoms, including 7 positive symptoms, 7 negative symptoms, and 16 general psychiatric symptoms. The severity of each symptom is rated on a scale ranging from 1 (minimal) to 7 (extreme); higher scores indicate increased symptomatology. Total PANSS scores include scores from all categories and range from 30 to 210 units on a scale.
Time Frame: 16 weeks (week 2 to week 18)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
score on a scale
  Wk 2 (Begin Treatment) PANSS Total Score | 81.0 (12.2) | 81.5 (13.0)
  Wk 18 (End Treatment) PANSS Total Score | 81.7 (13.3) | 79.7 (14.6)

2. Secondary Outcome: Change in MATRICS Consensus Cognitive Battery (MCCB) Overall Composite Scores From the Start to the End of the Study
Description: The MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia) Consensus Cognitive Battery (MCCB) is a standardized battery of 10 tests that measure 7 domains of cognitive performance: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. Overall composite t-scores are calculated using scores from all subtests. A t-score of 50 (10) is the mean (standard deviation) of the relevant reference population. Higher values indicate better performance.
Time Frame: 18 weeks (week 0 to week 18)
Measure: Mean (Standard Deviation); unit: t scores
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
t scores
  Wk 0 (Baseline) MCCB Score | 25.0 (12.0) | 19.5 (13.4)
  Wk 18 (End Treatment) MCCB Score | 26.8 (12.6) | 22.8 (13.6)

3. Secondary Outcome: Change in C-Reactive Protein From the Start to the End of the Study
Time Frame: 18 weeks (assessed at weeks 0, 10, and 18; weeks 0 and 18 reported)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
ng/ml
  CRP (Wk 0, Baseline) | 10402.8 (13488.2) | 8969.7 (9021.6)
  CRP (Wk 18, End Treatment) | 10198.5 (12110.9) | 10224.5 (13654.0)

4. Secondary Outcome: Change in Pentraxin-3 From the Start to the End of the Study
Time Frame: 18 weeks (assessed at weeks 0, 10, and 18; weeks 0 and 18 reported)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
ng/ml
  Pentraxin(Wk 0, Baseline) | 0.414 (0.534) | 0.461 (0.603)
  Pentraxin (Wk 18, End Treatment) | 0.394 (0.569) | 0.558 (0.695)

5. Secondary Outcome: Change in Anti-Saccharomyces Cerevisiae IgA Class Antibodies From the Start to the End of the Study
Time Frame: 18 weeks (assessed at weeks 0, 10, and 18; weeks 0 and 18 reported)
Measure: Mean (Standard Deviation); unit: units/ml
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
units/ml
  ASCA IGA (Wk 0, Baseline) | 0.195 (0.222) | 0.168 (0.163)
  ASCA IGA (Wk 18, End Treatment) | 0.226 (0.277) | 0.176 (0.184)

6. Secondary Outcome: Change in Interleukin-6 From the Start to the End of the Study
Time Frame: 18 weeks (assessed at weeks 0, 10, and 18; weeks 0 and 18 reported)
Measure: Mean (Standard Deviation); unit: pg/m
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
pg/m
  IL-6 (Wk 0, Baseline) | 0.623 (0.247) | 0.704 (0.478)
  IL-6 (Wk 18, End Treatment) | 0.694 (0.288) | 0.673 (0.357)

7. Secondary Outcome: Change in Tumor Necrosis Factor - Alpha From the Start to the End of the Study
Time Frame: 18 weeks (assessed at weeks 0, 10, and 18; weeks 0 and 18 reported)
Measure: Mean (Standard Deviation); unit: pg/m
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
pg/m
  TNF-a (Wk 0, Baseline) | 0.668 (0.393) | 0.538 (0.211)
  TNF-a (Wk 18, End Treatment) | 0.638 (0.362) | 0.520 (0.263)

8. Secondary Outcome: Change in Interferon Gamma From the Start to the End of the Study
Time Frame: 18 weeks (assessed at weeks 0, 10, and 18; weeks 0 and 18 reported)
Measure: Mean (Standard Deviation); unit: pg/m
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
Number analyzed (Participants) | 29 | 29
pg/m
  IFN-g (Wk 0, Baseline) | 0.514 (0.432) | 0.456 (0.172)
  IFN-g (Wk 18, End Treatment) | 0.478 (0.335) | 0.526 (0.222)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over an 18 week period, including the 2 week placebo run-in and the 16 week double-blind treatment phase.
Arm/Group | Sulforaphane Nutraceutical | Identical-appearing Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32 | 5/32
Other Adverse Events (participants affected / at risk) | 28/32 | 20/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulforaphane Nutraceutical (N=32) | Identical-appearing Placebo (N=32)
Schizophrenia exacerbation (Psychiatric disorders) | 2 (2) | 2 (3)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulforaphane Nutraceutical (N=32) | Identical-appearing Placebo (N=32)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 9 (9)
Cardiovascular symptoms (Cardiac disorders) | 1 (1) | 3 (3)
Gastrointestinal symptoms (Gastrointestinal disorders) | 12 (15) | 6 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Endocrine/metabolic symptoms (Endocrine disorders) | 4 (4) | 7 (8)
Dermatological symptoms (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Urinary symptoms (Renal and urinary disorders) | 2 (2) | 3 (3)
Psychiatric symptoms (Psychiatric disorders) | 11 (14) | 5 (11)
Hematological symptoms (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Other (General disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT02810964/Prot_SAP_000.pdf